CLINICAL TRIAL: NCT03760133
Title: The Change of Gut Microbiota After Bowel Preparation and the Effect of Probiotics: Randomized Controlled, Open-label Trial
Brief Title: The Change of Gut Microbiota After Bowel Preparation and the Effect of Probiotics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kosin University Gospel Hospital (Other)
Collaborators: Cell Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jae Hyun Kim, Assistant Professor, Kosin University Gospel Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-07-024
Record Dates: First submitted 2018-11-25; First posted 2018-11-30 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Gut Microbiota; Bowel Preparation; Colonoscopy
Keywords: Gut microbiota; Colonoscopy; Bowel preparation; Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- with Probiotics (Active Comparator): Participants included in this group will be taken probiotics for 1 month after bowel preparation for colonoscopy.
  Interventions: Drug: Duolac
- without Probiotics (No Intervention): Participants included in this group will not be taken probiotics for 1 month after bowel preparation for colonoscopy.

INTERVENTIONS:
Drug: Duolac — Participants included in this group will be taken probiotics for 1 month after bowel preparation for colonoscopy.
  Arms: with Probiotics

SUMMARY:
The purpose of this study is to investigate the relationship between the change of intestinal bacterial flora and the recovery, and the incidence of symptoms such as abdominal discomfort after colonoscopy. And the investigators will also analyze the effects of probiotics on the degree of change, recovery, and symptom development in intestinal flora.

DETAILED DESCRIPTION:
The investigators divided two groups. (total number = 100 subjects)

1. with probiotics group - 50 subjects

   * Participants included in this group will be taken probiotics for 1 month after bowel preparation for colonoscopy.
2. without probiotics group - 50 subjects

   * Participants included in this group will not be taken probiotics for 1 month after bowel preparation for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* adults between the age of 30 and 70

Exclusion Criteria:

* subjects with cancer or IBD (inflammatory bowel disease)
* subjects with history of abdominal surgery
* subjects who take medication related to gastrointestinal motility within 3 months
* subjects who take antibiotics within 3 months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The effect of probiotics on the change of gut microbiota after bowel preparation. | eight months
  Analysis the change of gut microbiota before and after bowel preparation for colonoscopy, and the effect of probiotics.

SECONDARY OUTCOMES:
The occurrence of symptoms | eight months
  Analysis the occurrence of symptoms including abdominal discomfort, diarrhea, constipation or abdominal blotting after bowel preparation for colonoscopy.
The correlation between symptoms and gut microbiota.. | eight months
  Analysis the the correlation between the symptoms after bowel preparation for colonoscopy and the changes of gut microbiota.

CONTACTS AND LOCATIONS:
Locations (1):
- Kosin University Gospel Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No
The investigators have no plan to share IPD to other researchers.